CLINICAL TRIAL: NCT04076839
Title: The Effectiveness of a Cognitive Training Program, Goal Management Training, on Reducing Cognitive Difficulties and Improving Every-day Functioning in Individuals With Affective Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Homewood Research Institute (Other)
Collaborators: McMaster University (Other); St. Joseph's Healthcare Hamilton (Other); Homewood Health Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-29
Record Dates: First submitted 2019-08-28; First posted 2019-09-03 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2019-08

CONDITIONS: Post-traumatic Stress Disorder; Cognitive Dysfunction
Keywords: cognitive remediation; public safety personnel; Goal Management Training; Group therapy; first responders; military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either: 1) a 9-week GMT program or 2) a 9-week wait-list control (WLC) condition. Participants will be tested at baseline prior to group commencement. Once the testing session is complete, the participants will be assigned to (GMT or WLC). Participants enrolled in the GMT program will attend 9-weeks of GMT sessions (2 hours/week for 9 weeks) and a post-intervention testing session date. Participants enrolled in the WLC group will be given a testing session date after 9 weeks has past. Participants will attend a final testing session (in 3 months' time; approximately 3 hours in duration). WLC will be offered a complimentary 9-week GMT program once the final testing session is complete. Following the completion of the complimentary 9-week GMT program, individuals in the WLC will complete post-intervention testing (1-2 weeks following the completion of GMT and again at 3 months, post GMT completion).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal Management Training (GMT) (Experimental): Goal Management Therapy is a structured, short-term, present-oriented cognitive remediation program with emphasis on mindfulness and practice in planning and completion of goal-oriented behaviors. The primary objective of GMT is to train patients to interrupt ongoing behavior through the resumption of executive control in order to define goal hierarchies and monitor performance in achieving goals. Sessions include instructional material, interactive tasks, discussion of patients' real-life deficits, and homework assignments. Participants assigned to this group will attend 9 weeks of GMT group sessions, each 2 hours in length, occurring once per week.
  Interventions: Behavioral: Goal Management Training
- Wait-list Control (No Intervention): Following baseline testing, participants randomly assigned to the wait-list control group will have no intervention during the 9 weeks that the GMT group attends their group sessions. Following the completion of the GMT group intervention, the wait-list control will attend a a testing session, and subsequently, a 3 month follow-up testing session, the results of which will be compared to those of the GMT group. This group will then be offered a complimentary 9-week GMT program once the final testing session is complete. Again, during these sessions participants will be required to complete questionnaires every third session in order to monitor their progress and symptoms. Following the completion of the complimentary 9-week GMT program, individuals in the WLC will complete post-intervention testing

INTERVENTIONS:
Behavioral: Goal Management Training — Goal Management Therapy is a structured, short-term, present-oriented cognitive remediation program with emphasis on mindfulness and practice in planning and completion of goal-oriented behaviors. The primary objective of GMT is to train patients to interrupt ongoing behavior through the resumption of executive control in order to define goal hierarchies and monitor performance in achieving goals. Sessions include instructional material, interactive tasks, discussion of patients' real-life deficits, and homework assignments.
  Arms: Goal Management Training (GMT)

SUMMARY:
This study investigates the utility of Goal Management Training (GMT) in patients with post-traumatic stress disorder (PTSD), in order to determine if this treatment is effective in improving cognitive function in patients with frontal-temporally mediated brain dysfunction. Specifically, the primary aim of this study is to examine whether a standardized 9-week program of GMT results in durable improvements in cognitive functioning relative to a wait-list control group. A secondary aim will be to determine whether participation in the GMT group is associated with long-term functional improvements. It is hypothesized that at post-treatment, participants with PTSD assigned to the GMT groups will show greater improvement in neuropsychological test performance and greater functional improvement compared to those in the wait-list group; these gains are expected to be maintained at 3 month follow-up.

DETAILED DESCRIPTION:
Given the potentially devastating impact of poor cognitive functioning on the ability of patients with PTSD to benefit from treatment interventions, and its association with poor functional outcomes, there is an urgent need to identify novel treatment interventions aimed at reducing cognitive dysfunction in these disorders. Accordingly, the aim of the present proposal is to conduct a randomized controlled trial among patients with PTSD, examining the efficacy of a well-established cognitive intervention (in the treatment of cognitive deficits), aimed at reducing attentional and executive dysfunction, known as Goal Management Training® (GMT) (See Levine et al., 2011). A secondary aim is to determine the longer-term impact of the GMT approach on functional outcomes.

The participants include 48 men and women with a primary diagnosis of with stable symptoms at the time of baseline assessment and reporting alterations in memory, attention, or executive functioning. Participants will be recruited from multiple sites: an inpatient post-traumatic stress recovery program in Ontario, Canada, and the program's external referral agencies that also service clients via outpatient services/ programs, external community agencies and support groups, and through social media.

Following determination of eligibility, participants will be randomly assigned, by using the randomized table of numbers method, to either: 1) a 9-week GMT program or 2) a 9-week wait-list control (WLC) condition (see Figure 1). Participants will be invited to attend a baseline testing session 1 prior to group commencement (approximately 4 hours in duration) where written consent will be obtained prior to any collection of data. Once the testing session is complete, the participants will be given information about what group they have been assigned to (GMT or WLC).

Participants enrolled in the GMT program attended the 9-week GMT sessions (2 hours/week for 9 weeks) and a post-intervention testing session date (1-2 weeks following the completion of the GMT; approximately 3 hours in duration). Participants enrolled in the WLC control group attended a testing session date after 9 weeks has past (approximately 3 hours in duration).

As each participant completed a post-intervention testing session (both GMT and WLC), they will be setup with the final testing session (in 3 months' time; approximately 3 hours in duration). WLC were offered a complimentary 9-week GMT program once the final testing session is complete. Following the completion of the complimentary 9-week GMT program, individuals in the WLC completed a post-intervention testing (1-2 weeks following the completion of GMT and again at 3 months, post GMT completion).

These data will be analyzed using 2 x 3 mixed-design split plot factorial ANCOVAs that treat Group (GMT vs. WLC) as a between-subjects factor and Time (baseline, post-intervention, 3 months; subjects nested within groups) as a within-subjects factor. In addition, within-subjects analyses of covariance (ANCOVAS) treating time (baseline, post-intervention, 3 months) as a within-subjects factor will be carried out on data collected from the GMT group and from the WLC group after they have completed the GMT arm of the study. PTSD symptom severity (CAPS), depressive symptom severity (BDI-II), severity of past trauma exposure (CTQ), and medication load, and additional psychological treatment (treatment information form) will serve as covariates in this model. Tukey's Honestly Significant Difference post-hoc test will be used for follow-up pair-wise comparisons of between-subjects' variables.

It is hypothesized that, post-treatment, participants with PTSD assigned to the GMT group will show significantly greater improvement in neuropsychological test performance and greater functional improvement compared to participants in the wait-list control group; these gains are expected to be maintained at 3-month-follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-70
* Are fluent in written and spoken English
* Are able to provide written informed consent
* Have a confirmed primary diagnosis of PTSD, history of PTSD diagnosis, or a history of trauma exposure as confirmed by the Mini International Neuropsychiatric Interview.

Exclusion Criteria:

* Are not current or former military personnel/ veterans or first responders/ public safety personnel
* Indicate alcohol and/or substance abuse within the past 3 months
* Have a recent history (within the past 12 months) of medical disorder known to adversely affect cognition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Change in score on Controlled Oral Word Association Task (COWAT) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  A neuropsychological assessment of verbal fluency, in which participants are asked to name as many words beginning with "F", "A", and "S" (Subscale: FAS). For each letter, they are given one minute to complete the task. Following this, the participant is required to name as many animals as they can within one minute (Subscale: Animals). Scores are calculated by adding unique words across FAS, and within Animals. These raw scores (i.e., FAS raw and Animals raw) are converted to scaled scores (i.e., FAS Scaled Score and Animals Scaled Score), which range between 0 and 19. The scaled scores are then converted to T scores (i.e., FAS T Score and Animals T Score), which range between 0 and 100. The T scores are corrected for sex, age, education, and ethnicity. Higher T scores indicate greater verbal fluency performance.
Change in score on Stroop Colour and Word Test | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  A neuropsychological assessment of processing speed (word and colour reading) and sensitivity to suppress habitual responses.The test produces the following scores: i) Word-Reading Score, which is the raw score that consists of the number of items completed in 45 seconds. ii) Colour-Naming Score, which is the raw score that consists of the number of items completed in 45 seconds. iii) Colour-Word Score, which is the raw score that consists of the number of items completed in 45 seconds, and iv) Interference Score, which is derived by subtracting a Predicted Colour-Word Score (obtained from the Stroop Manual) from the raw Colour-Word Score. Scores are then translated into T scores using a table obtained from the Stroop manual. Values for these T scores range between 3-98, and 21 and 80 for the Predicted Colour-Word Score. Overall, higher T scores indicate greater processing speed and ability to suppress habitual responses.
Change in score on Delis-Kaplan Executive Function System (D-KEFS) Tower Test | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  A neuropsychological assessment of planning, rule learning, response inhibition, and perseveration. Six scores are calculated: i) Total Achievement Score, which is the sum of achievement scores for all items administered. ii) Mean First-Move Time which reflects the average of the examinee's first move times. iii) Time-Per-Move Ratio, which indicates the average time the examinee takes to make each of his or her moves. iv) Move Accuracy Ratio is a means of assessing the efficiency with which the examinee constructed the towers. v) Total Rule Violations represents the total number of rule violations committed by the examinee across all items administered. vi) Rule-Violations-Per-Item Ratio, reflects the average number of rule violations made by the examinee relative to the number of items administered. The total number of rule violations across all items administered is divided by the number of items administered. Higher scores indicate greater executive functioning performance.
Change in score on Trail Making Test Part A & B (TMT A & TMT B) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  A neuropsychological assessment in which participants are required to sequence two stimulus sets while alternating between them. Scoring is expressed in terms of the time in seconds required for completion of each of the two parts of the test (i.e., TMT A and TMT B). The raw scores for each part of the test are translated to scaled scores (i.e., TMT A Scaled Score and TMT B Scaled Score) and scaled scores may range between 0 and 19. The scaled scores are then translated to T scores (i.e., TMT A T Score and TMT B T Score) corrected for sex, age, education, and ethnicity. The T scores may range between 0 and 100. Individuals with higher T scores indicate better attention, mental flexibility, and speed in comparison to those with lower T scores.
Change in score on Wechsler Adult Intelligence Scale-IV (WAIS-IV), Coding Subtest | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  A neuropsychological assessment of processing speed. In a time limit of 120 seconds, the participant copies symbols that are paired with numbers based on a symbol key. The total raw score is calculated by scoring 1 point for each correctly drawn symbol completed within the time limit. Raw scores range between 0 and 135 points. The raw score is converted to a scaled score corrected for age and the scaled score may range between 1 and 19. Higher scaled scores indicate greater processing speed than lower scaled scores.
Change in score on Conners Continuous Performance Task Third Edition (CPT-III) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  A neuropsychological assessment of inattentiveness, impulsivity, sustained attention, and vigilance. Values include: i) D-prime-discrimination of non targets from targets; ii) Omissions- all missed targets; iii) Commissions- all incorrect responses to non-targets; iv) Perseverations- response in less than 100 milliseconds following the presentation of a stimulus; v) Hit Reaction Time- mean response speed measured in milliseconds for all non-perseverative responses made during the entire administration; vi) Hit Reaction Time SD-consistency of response speed to targets for the entire administration; vii) Variability- response speed consistency; viii) Hit Reaction Time Block Change- slope of change in Hit Reaction Time across the six blocks of the administration; and ix) Hit Reaction Time Inter-Stimulus Interval Change- slope of change in reaction time across the three inter-stimulus intervals. All scores are presented in T scores with higher T scores indicating worse performance.
Change in score on California Verbal Learning Test II (CVLT-II) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  A word list neuropsychological assessment, which provides indices of immediate and delayed memory performance, interference learning, and recognition. Software is utilized to score the CVLT-II, which computes all raw scores and standardized scores, corrected for the examinee's age and gender. Values of interest within the study include: i) Level of Immediate Recall; ii) Level of Delayed Recall, iii)Learning Characteristics, iv) Recall Errors, and v) Delayed Recognition Trials. In general, higher standard scores indicate intact performance; however, in other cases (e.g., Recall Errors) higher standard scores reflect greater deficits.
Change in score on Rivermead Behavioural Memory Test Second Edition (RBMT-II) Prospective Memory Tasks | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  Participants will be asked to complete two prospective memory tasks (Belongings and Appointments) where they will be given specific instructions and asked to independently act on these instructions at specific time points throughout the testing. Raw scores for Belongings and Appointments will be assessed. The raw score for Belongings may range between 0 and 8, while the raw score for Appointments may range between 0 and 4. Higher raw scores indicate better recall.
Wechsler Abbreviated Scale of Intelligence - II (WASI-II): Vocabulary and Matrix Reasoning Subtests | Administered to GMT participants and Waitlist Participants only at baseline.
  The WASI-II is a brief neuropsychological assessment aimed to provide an estimate of current intellectual functioning. The two-subtest form of the WASI-II consists of Vocabulary and Matrix Reasoning and provides a Full Scale IQ (FSIQ-2). In the Vocabulary subtest, participants give oral definitions for words (total raw scores may range between 0 and 59). For Matrix Reasoning, the participant looks at a matrix with a section missing and identifies the missing section by pointing to or stating the number of their response (total raw scores may range between 0 and 30). The subtests' total raw scores are converted to age-corrected T scores (T scores may range between 20 and 80 for each subtest). The FSIQ-2 is the sum of T scores on Vocabulary and Matrix Reasoning. FSIQ-2 scores may range between 45 and 160, with higher FSIQ-2 scores indicating higher intelligence.
Wechsler Test of Adult Reading (WTAR) | Administered to GMT participants and Waitlist Participants only at baseline.
  The WTAR assesses premorbid intellectual functioning in adults. The WTAR requires the participant to read out loud irregularly spelled words. The raw score ranges between 0 and 50. The WTAR raw score is converted to a standard score and the standard score may range between 50 and 134. Intelligence scores are also predicted by WTAR performance and demographics and intelligence scores may range between 89 and 118. Higher intelligence scores indicate greater premorbid intellectual functioning.
Change in Score on Multidimensional Scale of Independent Functioning (MSIF) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  A semi-structured interview assessing participant report of i) work (e.g., competitive, supported, dependent care, volunteer); ii) education (e.g., college, vocational, certificate school, rehabilitation training program); and iii) residential activities (e.g., where the participant is living, what responsibilities the participant has). Each domain (i.e., work, education, and residential activities) is assessed according to role position, support, and performance. Scores for these areas may range between 1 and 7, with higher values indicating greater impairment in functioning. Furthermore, a global rating for role position, support, performance, and overall functioning is given. Scores for the global ratings also may range from 1 to 7, with higher values indicating greater impairment in functioning.
Change in Score on World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The WHODAS 2.0 is a 12-item self-report measure of six functional domains, including cognition, mobility, self-care, getting along with others, life activities, and participation in the community. The WHODAS 2.0 uses a Likert scale ranging from 0 ("No difficulty") to 4 ("Extreme difficulty or cannot do"). Values across the 12 items are summed, with the total score ranging between 0 and 48. Higher values indicate greater functional impairment.
Change in Score on Sheehan Disability Scale (SDS) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The SDS is a 3-item self-report measure of disability in work, social relationships, and family life. The three items, which are scored on a Likert scale between 0 and 10, are summed into a single dimensional measure of global functional impairment. The SDS total score may range from 0 to 30, with higher scores indicating greater impairment.
Change in Score on Goal Attainment Scaling (GAS) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  Description: The GAS is a method for defining individual participant goals and the standardized measurement of progress towards these goals. Overall goal attainment is transformed into a T score, with higher T scores indicating greater goal attainment.
Change in Score on Cognitive Failures Questionnaire (CFQ) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months). Also GMT sessions 1,3,6, and 9
  The CFQ is a 25-item self-report measure that captures daily errors in distractibility, blunders, names, and memory. Each item is rated on a Likert scale from 0 ("Never") to 4 ("Very often"). The CFQ has four subscales that include: i) Memory (i.e., sum of scores on items 16, 18, 12, 17, 23, 13, 6, 3 for a total score between 0 and 32); ii) Distractibility (i.e., sum of scores on items 1, 15, 2, 19, 21, 22, 3, 4, 25 for a total score between 0 and 36); iii) Blunders (i.e., sum of scores on items 9, 8, 10, 24, 5, 14, 11 for a total score between 0 and 28); and iv) Names (i.e., sum of scores on items 20 and 7 for a total score between 0 and 8). The CFQ total score is the sum of the 25 items, with total values ranging between 0 and 100. Higher scores indicate greater self-reported impairment in cognitive functioning.
Change in Score on Dysexecutive Questionnaire (DEX) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The DEX is a 20-item self-report measure that asks participants to rate inhibition, positive and negative affect, memory, and intention. Each item is rated on a Likert scale from 0 ("Never") to 4 ("Very often"). The DEX Total score is the sum of all items and the total score may range from 0 to 80. Higher scores indicate greater self-reported cognitive impairment.

SECONDARY OUTCOMES:
Demographic Information | Administered to GMT participants and Waitlist Participants only at baseline.
  Description: A self-report measure assessing demographic information including age, sex, race, education, marital status, employment status, and employment type (e.g., active military member, veteran, public safety personnel, first responder, or other).
Mini International Neuropsychiatric Interview 7.0 (M.I.N.I.) | Administered to GMT participants and Waitlist Participants only at baseline.
  Description: The M.I.N.I. is a structured clinician administered interview in order to assess psychiatric disorders according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition. The M.I.N.I. is divided into modules identified by letters, each corresponding to a diagnostic module. At the end of each module, diagnostic boxes permit the clinician to indicate whether diagnostic criteria are met. The diagnostic modules utilized within the study include: i) Major Depressive Episode; ii) Suicidality; iii)Manic and Hypomanic Episodes; iv)Panic Disorder; v) Agoraphobia; vi)Social Anxiety Disorder; vii)Obsessive Compulsive Disorder; viii) Alcohol Use Disorder; ix)Substance Use Disorder; x)Psychotic Disorders and Mood Disorder with Psychotic Features; xi)Anorexia Nervosa; xii)Bulimia Nervosa; xiii)Binge Eating Disorder; and xiiii)Generalized Anxiety Disorder.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Administered to GMT participants and Waitlist Participants only at baseline.
  The CAPS-5 is a semi-structured interview that assesses the DSM-5's PTSD diagnostic criteria in the past month. In order to meet the diagnostic criteria for PTSD, individuals must indicate an index trauma and have at least one intrusion symptom, an avoidance symptom, two cognition and mood symptoms, and two arousal and reactivity symptoms. Further, the duration of the symptoms must be present for at least one month and must cause either distress or impairment in functioning. Total scores on the CAPS-5 for severity may range between 0 and 80, with higher scores indicating greater symptom severity.
Life Events Checklist for DSM-5 (LEC) | Administered to GMT participants and Waitlist Participants only at baseline.
  The LEC is a self-report measure, which probes exposure to common traumatic events over the lifespan (e.g., natural disasters, sexual violence, violence, etc.). There is no formal scoring protocol or interpretation per se, other than identifying whether a person has experienced one or more of the events listed.
Childhood Trauma Questionnaire (CTQ) | Administered to GMT participants and Waitlist Participants only at baseline.
  A self-report measure, which assesses for exposure to five forms of common childhood trauma (i.e., sexual abuse, physical abuse, emotional abuse, physical neglect, emotional neglect). Each item is rated on a Likert scale from 1 ("Never true") to 5 ("Very often true"). All subscales (i.e., the five forms of childhood trauma) have a possible score range of 5 to 25.
Change in Score on Psychological Treatment and Medication Assessment | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  A clinician administered interview assessing examinee participation in any psychological treatment (e.g., cognitive behavioural therapy) outside of the study and medications prescribed throughout the course of the study.
Change in Score on PTSD Checklist for DSM-5 (PCL-5) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months). Also GMT sessions 1,3,6, and 9
  The PCL-5 is a 20-item self-report measure, which assesses the severity of PTSD symptoms according to the diagnostic criteria outlined in the DSM-5. The symptom domains include intrusions (items 1 through 5; scores summed for a total between 0 and 20), avoidance (items 6 through 7; scores summed for a total between 0 and 8), negative alterations in mood and cognitions (items 8 through 14; scores summed for a total between 0 and 28), and alterations in arousal and reactivity (items 15 through 20; scores summed for a total between 0 and 24). Participants rate the severity of their symptoms in the past month on a Likert scale from 0 ("Not at all") to 4 ("Extremely"). A total PCL-5 score is derived by summing all the values of the items and the total score may range between 0 and 80. A cut-point of 33 is suggested to indicate a probable PTSD diagnosis.
Change in Score on Multiscale Dissociation Inventory (MDI) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months). Also GMT sessions 1,3,6, and 9
  The MDI is a 30-item self-report measure, which assesses six domains of dissociative symptoms over the past month, including disengagement (items 1, 7, 13, 19, 25; scores summed for a total between 5 and 25), depersonalization (items 2, 8, 14, 20, 26; scores summed for a total between 5 and 25), derealization (items 3, 9, 15, 21, 27; scores summed for a total between 5 and 25), emotional constriction (items 4, 10, 16, 22, 28; scores summed for a total between 5 and 35), memory disturbance (items 5, 11,17,23,29; scores summed for a total between 5 and 25), and identity dissociation (items 6, 12, 18, 24, 30; scores summed for a total between 5 and 25). Participants rate the severity of their symptoms within the last month on a Likert scale from 1 ("Never") to 5 ("Very often"). A total MDI score is derived by summing all the values of the items and the total score may range between 30 and 150. Higher total scores indicate greater dissociation.
Change in Score on Difficulties in Emotion Regulation Scale (DERS) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months). Also GMT sessions 1,3,6, and 9
  The DERS is a 36-item self-report measure, which assesses difficulties with emotion regulation across six domains including nonacceptance of emotional responses (items 11, 12, 21, 23, 25, 29; scores summed for a total between 6 and 30), difficulty engaging in goal-directed behavior (items 13, 18, 20, 26, 33; scores summed for a total between 5 and 25), impulse control difficulties (items 3, 14, 19, 24, 27, 32; scores summed for a total between 6 and 30), lack of emotional awareness (items 2, 6, 8, 10, 17, 34; scores summed for a total between 6 and 30), limited access to emotion regulation strategies (items 15, 16, 22, 28, 30, 31, 35, 36; scores summed for a total between 8 and 40), and lack of emotional clarity (items 1, 4, 5, 7, 9; scores summed for a total between 5 and 25). A total DERS score is derived by summing all the values of the items and this score may range between 36 and 180. Higher scores indicate greater dysfunction with emotion regulation.
Change in Score on Beck Depression Inventory II (BDI-II) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months). Also GMT sessions 1,3,6, and 9
  The BDI-II is a 21-item self-report questionnaire that assesses the presence and severity of symptoms of depression over the past month. Respondents rate their symptoms on a Likert scale from 0 to 3. A total BDI-II score is derived by summing all the values of the items and the total score may range between 0 and 63. Higher scores reflect greater depression symptom severity.
Change in Score on Beck Anxiety Inventory (BAI) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months). Also GMT sessions 1,3,6, and 9
  The BAI is a 21-item self-report questionnaire that assesses anxiety symptoms over the past month. Participants rate their symptoms on a Likert scale from 0 ("Not at all") to 3 ("Severely - it bothered me a lot"). A total BAI score is derived by summing all the values of the items and the total score may range between 0 and 63. Higher scores indicate greater anxiety symptom severity.
Change in Score on Emotion Regulation Questionnaire (ERQ) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The ERQ is a 10-item self-report assessment that is designed to assess individual differences in the habitual use of cognitive reappraisal and expressive suppression. Each of the items is scored on a Likert scale from 1 ("Strongly disagree") to 7 ("Strongly agree"). Scoring for the Cognitive Reappraisal subscale includes items 1, 3, 5, 7, 8, and 10 and scores are summed for totals ranging between 6 and 42. Here, higher scores indicate greater use of cognitive reappraisal. Scoring for the Expressive Suppression subscale includes items 2, 4, 6, and 9, and scores are summed for totals ranging between 4 and 28. Here, higher scores indicate greater use of expressive suppression.
Change in Score on Toronto Alexithymia Scale (TAS) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The TAS is a 20-item self-report measure, which assesses difficulties recognizing and naming emotions across three domains including, difficulty identifying feelings (items 1, 3, 6, 7,9, 13, 14; scores summed for a total between 7 and 35), difficulty describing feelings(items 2, 4, 11, 12, 17; scores summed for a total between 5 and 25), and externally-oriented thinking (items 5, 8, 10, 15, 16, 18, 19, 20; scores summed for a total between 8 and 40). A total TAS score is derived by summing all the values of the items and the total score may range between 20 and 100. Individuals with scores less than or equal to 51 are interpreted as having no alexithymia. Further, individuals with scores between 52 and 60 are interpreted as having possible alexithymia. Finally, individuals with scores greater than or equal to 61 are interpreted as having alexithymia.
Change in Score on Dissociation Tension Scale (DSS) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The DSS is a self-report measure, which assesses the psychological and somatoform dissociative features as well as aversive inner tension occurring within the past 7 days. The DSS contains 21 items assessing dissociative symptoms and 1 additional item assessing aversive inner tension. Ratings are made on a time-oriented scale ranging from 0% ("Never") to 100% ("Constantly"). A total DSS score is derived by summing the values of the 21-items and the total score may range between 0 and 2100. Higher scores indicate greater dissociative symptoms.
Change in Score on The Short Version of the Borderline Symptom List (BSL-23) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The BSL-23 is a self-report measure, which assesses for the presence of borderline-typical symptomatology in the past week. It contains 23 items that assess borderline-typical symptomatology (items are rated on a Likert scale between 0 ("Not at all") and 4 ("Very strong"); scores summed for a total between 0 and 92), an item asking participants to rate the quality of their overall personal state in the past week (item is rated on a Likert scale between 0% ("Very bad") and 100% ("Excellent")), and 11 supplemental items assessing the frequency of risk behaviors within the past week (items are rated on a Likert scale between 0 ("Not at all") and 4 ("Daily or more often"); scores may be summed for a total between 0 and 44). The total score of the BSL-23 is calculated by dividing the total sum of the 23 items by the number of items (i.e., the total BSL-23 score may range from 0.0 to 4.0), with an average of 2 or greater suggestive of a diagnosis of borderline personality disorder.
Change in Score on Moral Injury Events Scale (MIES) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The MIES is a 9-item self-report measure assessing moral injury along two dimensions in military and veteran populations - perceived transgressions and perceived betrayals. Each item is rated on a Likert scale from 1 ("Strongly disagree") to 6 ("Strongly agree"). The Perceived Transgressions subscale consists of the items 1 through 6 (scores summed for a total between 6 and 36), while the Perceived Betrayals subscale consists of the items 7 through 9 (scores summed for a total between 3 and 18). The total MIES score is the sum of all 9 items, with a total score ranging between 9 and 54. Higher values on the subscales and total score indicate greater moral injury.
Change in Score on Trauma-Related Guilt Inventory (TRGI) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The TRGI is a self-report measure that assesses common experiences of guilt for trauma survivors, consisting of six subscales: i) Global Guilt Scale (sum of scores on Items 13, 18, 22, 25 divided by 4; ii) Distress Scale (sum of scores on Items 2, 6, 10, 15, 20, 24 divided by 6; iii) Guilt Cognitions Scale (sum of scores on Items 1, 3-5, 7-9, 11, 12, 14, 16, 17, 19, 21, 23, 26-32 divided by 22; iv)Hindsight-Bias/Responsibility Subscale (sum of scores on Items 1, 5, 9, 14, 19, 23, 26 divided by 7; v)Wrongdoing Subscale (sum of scores on Items 3, 7, 11, 16, 21 divided by 5; and vi) Lack of Justification Subscale (sum of scores on Items 4, 8, 12, 17 divided by 4. Mean score on each scale may range between 0 and 4. Each item is rated on a Likert scale from 0 ("Never") to 4 ("Always"). Higher values on the subscales indicate greater difficulties with trauma-related guilt.
Change in Score on Trauma-Related Shame Inventory (TRSI) | GMT group: Baseline, post-treatment (9 weeks), and 3 months. Wait list control: Baseline, post 9 week delay period, post 3 month delay period, post GMT (8 months), 3 months post-treatment (11 months)
  The TRSI is a 24-item self-report measure assessing shame related to traumatic experiences across four subscales: i) Internal-Referenced Shame - Condemnation (items 1,5,10,13,15,21; scores summed for a total between 0 and 18); ii) Internal-Referenced Shame - Affective-Behavioural (items 3,8,9,11,20,23; scores summed for a total between 0 and 18); iii) External-Referenced Shame - Condemnation (items 12,17,2,4,6,14; scores summed for a total between 0 and18); and iv) External-Referenced Shame - Affective-Behavioural (items 16,19,24,22,18,7; scores summed for a total between 0 and 18). Each item is assessed on a Likert scale from 0 ("Not true of me") to 3 ("Completely true of me"). The total TRSI score is the sum of all 24 items, with a total score ranging between 0 and 72. Higher values on the subscales and total score indicate greater difficulties with trauma-related shame.
GMT Treatment Evaluation Form | Anonymous feedback collected following the participation in the GMT treatment portion of the study (9 weeks for GMT group, 8 months for wait list control)
  An anonymous form requesting participants to provide an evaluation of their experience in the GMT groups.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McKinnon, PhD, Principal Investigator — McMaster University, Homewood Research Institute
Locations (1):
- Homewood Research Institute, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aupperle RL, Melrose AJ, Stein MB, Paulus MP. Executive function and PTSD: disengaging from trauma. Neuropharmacology. 2012 Feb;62(2):686-94. doi: 10.1016/j.neuropharm.2011.02.008. Epub 2011 Feb 22. PMID 21349277
- [Background] Levine B, Robertson IH, Clare L, Carter G, Hong J, Wilson BA, Duncan J, Stuss DT. Rehabilitation of executive functioning: an experimental-clinical validation of goal management training. J Int Neuropsychol Soc. 2000 Mar;6(3):299-312. doi: 10.1017/s1355617700633052. PMID 10824502
- [Background] Polak AR, Witteveen AB, Reitsma JB, Olff M. The role of executive function in posttraumatic stress disorder: a systematic review. J Affect Disord. 2012 Dec 1;141(1):11-21. doi: 10.1016/j.jad.2012.01.001. Epub 2012 Feb 5. PMID 22310036
- [Background] Rockwood K, Joyce B, Stolee P. Use of goal attainment scaling in measuring clinically important change in cognitive rehabilitation patients. J Clin Epidemiol. 1997 May;50(5):581-8. doi: 10.1016/s0895-4356(97)00014-0. PMID 9180650
- [Background] Saunders N, Downham R, Turman B, Kropotov J, Clark R, Yumash R, Szatmary A. Working memory training with tDCS improves behavioral and neurophysiological symptoms in pilot group with post-traumatic stress disorder (PTSD) and with poor working memory. Neurocase. 2015;21(3):271-8. doi: 10.1080/13554794.2014.890727. Epub 2014 Feb 28. PMID 24579831